CLINICAL TRIAL: NCT01759849
Title: Effect of in Vitro Blocking the Common Beta Chain on the Function of Blood, Bone Marrow and Sputum Cells Collected From Asthmatic Donors.
Brief Title: Effect of in Vitro Blocking the Common Beta Chain on Cell Viability in Asthma
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: CSL Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: Bc in vitro study
Record Dates: First submitted 2012-12-17; First posted 2013-01-03 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Asthma
Keywords: Asthma; β-chain signaling; allergen inhalation challenges; sputum; bone marrow aspirate; blood collection; -methacholine challenge
MeSH Terms: conditions — Asthma | interventions — Allergens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, bone marrow and induced sputum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allergen challenge: Determination of the effects of a β-chain monoclonal antibody (MAb) on the function of cells naturally activated by in vivo allergen exposure, from donors with allergen-induced asthma
  Interventions: Other: Allergen

INTERVENTIONS:
Other: Allergen — Allergen extract is administered by inhalation.

SUMMARY:
This study examines in vitro blockade of signaling through the β-chain, on viability, activation and differentiation of eosinophils and their progenitors collected in sputum, blood and bone marrow samples pre and post-allergen challenge from mild atopic asthmatic subjects.

DETAILED DESCRIPTION:
The experiments will use sputum samples induced from subjects with mild asthma, undergoing allergen inhalation challenges. In general, each sample will be composed of >10% neutrophils and >10% macrophages. Samples collected pre-allergen will have a low frequency of eosinophils and lymphocytes (<1%), however the percentage of eosinophils will increase to approximately 12% following allergen challenges. The sputum samples will be processed in DPBS (without dithiothreitol), and the cell suspension will be adjusted to 1 million cells/ml in DMEM with penicillin and streptomycin. A cytospin will be made for differential cell counts. The mixed cell population at 5 million cells/ml will be incubated for 48 hours at 37 degrees Celcius ± β-chain MAb at a concentration of 100 mcg/ml. After 48 hours the cell culture medium will be removed for assay of cytokines and chemokines by ELISA. Cells will be resuspended in PBS and Binding Buffer (BD Pharmingen, Cat no. 556454),stained for assessments by flow cytometry, and analyzed in duplicate.

Experiments will use blood (80 ml) and bone marrow aspirates (5ml) from atopic asthmatics taken pre and 24hr post allergen challenge. Methylcult micro-culture colonogenic assays will be performed to enumerate outgrowth of Eo/Baso-CFU and GM-CFU from CD34+ cells populations collected from the blood and bone marrow samples. Methylcult assays will be performed with CD34+ enriched cell populations in the presence of IL-5,IL-3 and GM-CSF +/- CSL311. Following 14 days culture, colonies will be enumerated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers 18 through 65 years of age.
* General good health
* Mild to moderate, stable, allergic asthma
* History of episodic wheeze and shortness of breath; FEV1 at baseline at least 70% of the predicted value
* Able to understand and give written informed consent and has signed a written informed consent form approved by the investigator's REB
* Positive methacholine challenge
* Positive skin-prick test to common aeroallergens (including cat, dust mite, grass, pollen)
* Positive allergen-induced airway bronchoconstriction (a fall in FEV1 of at least 20% from baseline)

Exclusion Criteria:

* A worsening of asthma or a respiratory tract infection within 6 weeks preceding study entry
* Use of corticosteroids, immunosuppressives, anticoagulants (warfarin or heparin) within 28 days prior to randomization into the study
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs) within 48 hours of dosing or aspirin with 7 days of dosing
* Have chronic use of any other medication for treatment of allergic lung disease other than short- and intermediate-acting ß2-agonists or ipratropium bromide
* Use of caffeine-containing products or medications for 12 hours or alcohol or over the counter drugs including aspirin, cold and allergy medications for 48 hours or inhaled bronchodilators for 8 hours prior to methacholine and allergen challenges
* Use of tobacco products of any kind currently or within the previous 12 months, or smoking history > 10 pack years.
* Lung disease other than mild to moderate allergic asthma
* Unwillingness or inability to comply with the study protocol for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with mild allergic asthma.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Sputum Collection | 7 hours post allergen
  Three baseline sample collections will ensure sufficient numbers of cells are collected for proposed outcomes. Post allergen cells will be examined at time points when these populations are known to be at their highest frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Gail M Gauvreau, PhD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- McMaster University Medical Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study publication — https://www.ncbi.nlm.nih.gov/pubmed/26651396